CLINICAL TRIAL: NCT04389268
Title: Predictive Value of P300 Event-related Potential Component in Early Cognitive Impairment in Patients With Uncomplicated Newly Diagnosed Hepatitis C Virus
Brief Title: P300 in Early Cognitive Impairment in Hepatitis C Virus
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University HCV
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Hepatitis C; Cognitive Impairment
Keywords: Hepatitis C, Cognitive Impairment
MeSH Terms: conditions — Hepatitis C; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCV patients: Patients with uncomplicated newly diagnosed hepatitis C virus
  Interventions: Diagnostic Test: Visual Event-Related Potentials
- Control group: Age and sex matched with patients
  Interventions: Diagnostic Test: Visual Event-Related Potentials

INTERVENTIONS:
Diagnostic Test: Visual Event-Related Potentials — Auditory P300-evoked brain potential: an eventrelated potential of cognitive neurophysiological significance. It represents the brain response to certain sensory/cognitive stimuli by paying attention to the different stimulus among the stereotypical ones (the auditory oddball paradigm). It measures mainly the decision-making process (Polich and Kok, 1995).

SUMMARY:
Approximately 50% of patients with hepatitis C have complaints of fatigue and cognitive deficits even before the development of significant hepatic impairment.

DETAILED DESCRIPTION:
Assessing the influence of HCV infection on the development of cognitive changes involves many challenges. The frequent presence of confounding factors such as illicit drug use, depression, and cirrhosis has the potential to produce cognitive impairment and therefore obscuring the role of HCV infection as a major actor in the development of cognitive impairment.

The presence of brain dysfunction in patients with liver cirrhosis is well known. Zeegen et al. described in 1970, through the use of neuropsychological tests, the occurrence of cognitive changes involving mainly psychomotor speed, attention, and executive function in cirrhotics who did not have clinical criteria for hepatic encephalopathy. This condition is currently called minimal hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed HCV infection

Exclusion Criteria:

* Any neuropsychiatric disease that cause impaired cognition

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 100 participants consisted of 50 HCV patients and 50 healthy control, age and sex matched.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Auditory P300-evoked brain potential | 24-72 hours
  Auditory P300-evoked brain potential: an eventrelated potential of cognitive neurophysiological significance. It represents the brain response to certain sensory/cognitive stimuli by paying attention to the different stimulus among the stereotypical ones (the auditory oddball paradigm). It measures mainly the decision-making process (Polich and Kok, 1995).

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Latt NL. Update on the Management of Hepatitis C Virus Infection in the Setting of Chronic Kidney Disease and Kidney Transplantation. Gastroenterol Hepatol (N Y). 2018 Dec;14(12):687-705. PMID 30804716
- [Background] Louie KS, St Laurent S, Forssen UM, Mundy LM, Pimenta JM. The high comorbidity burden of the hepatitis C virus infected population in the United States. BMC Infect Dis. 2012 Apr 11;12:86. doi: 10.1186/1471-2334-12-86. PMID 22494445
- [Background] Barreira DP, Marinho RT, Bicho M, Fialho R, Ouakinin SRS. Psychosocial and Neurocognitive Factors Associated With Hepatitis C - Implications for Future Health and Wellbeing. Front Psychol. 2019 Jan 9;9:2666. doi: 10.3389/fpsyg.2018.02666. eCollection 2018. PMID 30687151
- [Background] Polaris Observatory HCV Collaborators. Global prevalence and genotype distribution of hepatitis C virus infection in 2015: a modelling study. Lancet Gastroenterol Hepatol. 2017 Mar;2(3):161-176. doi: 10.1016/S2468-1253(16)30181-9. Epub 2016 Dec 16. PMID 28404132
- [Background] Waked I, Doss W, El-Sayed MH, Estes C, Razavi H, Shiha G, Yosry A, Esmat G. The current and future disease burden of chronic hepatitis C virus infection in Egypt. Arab J Gastroenterol. 2014 Jun;15(2):45-52. doi: 10.1016/j.ajg.2014.04.003. Epub 2014 Jun 6. No abstract available. PMID 25097045